CLINICAL TRIAL: NCT03782714
Title: Clinical and Radiographic Evaluation of Low-level Laser Therapy in Human Primary Molar Pulpotomies: A Randomized Controlled Clinical Trial
Brief Title: Low-level Laser Therapy Versus Formocresol in Primary Molar Pulpotomies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Najlaa Alamoudi, Professor at the Pediatric Dentistry Department, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Alaa Nadhreen
Record Dates: First submitted 2018-12-16; First posted 2018-12-20 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Pulpotomy
Keywords: Low-level laser therapy, pulpotomy, formocresol
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: It is a split-mouth randomized controlled clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low-level laser therapy group (Experimental): This group of teeth received laser irradiation after amputation of coronal pulp
  Interventions: Device: Low-level laser therapy
- Formocresol group (No Intervention): This group of teeth received the gold standard medication (formocresol) after coronal pulp amputation

INTERVENTIONS:
Device: Low-level laser therapy — It is a diode laser device that has laser set at low level, used for pain relief and inflammation reduction to induce healing
  Arms: Low-level laser therapy group

SUMMARY:
This study aimed to assess and compare the clinical and radiographic success rates of LLLT and FC for pulpotomy in human primary teeth. One hundred and six primary molars from 36 children aging five to eight years were included and randomly assigned into two equal groups; LLLT group and FC group. Teeth were evaluated clinically and radiographically at 3, 6 and 12 months.

DETAILED DESCRIPTION:
Background: Various agents are available to dress the remaining pulp tissue after pulpotomy procedure with the formocresol (FC) being the gold standard for the last 60 years. Nowadays, low-level laser therapy (LLLT) becomes a technique of interest, due to its many characteristics. However, the literature available on its success in pulpotomy is limited and reported conflicting results.

Aim of the study: To assess and compare the clinical and radiographic success rates of LLLT and FC for pulpotomy in human primary teeth.

Materials and methods: Utilizing split-mouth technique, the sample consisted of 106 primary molars from 36 children aging five to eight years. The teeth were selected based on specific clinical and radiographic inclusion criteria and randomly assigned into two equal groups; LLLT group and FC group. All the 106 primary molars were indicated for pulpotomy, where 53 teeth were treated using FC and 53 teeth were treated with LLLT. Teeth were evaluated clinically and radiographically at 3, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

Children inclusion criteria:

* Children aged 5-8 years with at least two bilateral deep carious primary molars indicated for pulpotomy.
* Children who are physically and mentally healthy without any known medical history of systemic conditions contraindicating pulp therapy.
* Children who had "positive" or "definitely positive" behavioral ratings according to the Frankl behavior classification scale (Frankl, 1962).
* Children whose parents signed an informed consent for the child's participation in the study.

Teeth inclusion criteria:

Teeth were selected according to clinical and radiographic criteria.

Clinically, the study included:

* Teeth with restorable crowns
* Teeth with pathologic carious exposure of vital pulps
* Teeth with no tenderness to percussion, physiologic or pathologic mobility or any clinical evidence of pulp inflammation or degeneration such as history of swelling, pain or presence of sinus tract.

Radiographically, the recruited teeth should have:

* Normal radiographic appearance with healthy supporting tissues
* No pulp calcification
* No internal or external root resorption
* No periapical or inter-radicular radiolucency
* At least two thirds of the root remaining (not more than one third of the root is physiologically resorbed)

Exclusion Criteria:

* Any child complained of clinical signs such as pain, swelling, abnormal mobility, vertical or lateral tenderness to percussion was excluded from the study.
* Radiographically, any child with signs of internal or external root resorption or periapical or inter-radicular pathology was omitted from the study.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Clinical success rate | 3 months
  The pulpotomy procedure was considered clinically successful if there were no pain, swelling, tenderness to percussion, abscess or abnormal mobility
Clinical success rate | 6 months
  The pulpotomy procedure was considered clinically successful if there were no pain, swelling, tenderness to percussion, abscess or abnormal mobility
Clinical success rate | 12 months
  The pulpotomy procedure was considered clinically successful if there were no pain, swelling, tenderness to percussion, abscess or abnormal mobility
Radiographic success rate | 3 months
  The pulpotomy procedure was considered clinically successful if it demonstrated the following criteria:
  1. Normal periodontal ligament space
  2. No inter-radicular or periapical radiolucency
  3. No internal or external root resorption
Radiographic success rate | 6 months
  The pulpotomy procedure was considered clinically successful if it demonstrated the following criteria:
  1. Normal periodontal ligament space
  2. No inter-radicular or periapical radiolucency
  3. No internal or external root resorption
Radiographic success rate | 12 months
  The pulpotomy procedure was considered clinically successful if it demonstrated the following criteria:
  1. Normal periodontal ligament space
  2. No inter-radicular or periapical radiolucency
  3. No internal or external root resorption

CONTACTS AND LOCATIONS:
Locations (1):
- King Abdulaziz University, Dental University Hospital, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No